CLINICAL TRIAL: NCT05576207
Title: Balanced Energy and Protein (BEP) Supplementation Research in Bangladesh (JiVitA-BEP IR)
Brief Title: BEP Supplementation Research in Bangladesh (JiVitA-BEP-IR)
Acronym: Target-BEP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); BRAC James P Grant School of Public Health, BRAC University (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: INV-033381; IRB00021021 (Other: JHSPH IRB)
Record Dates: First submitted 2022-10-05; First posted 2022-10-12 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Fetal Growth Retardation; Low Birth Weight; Preterm Birth; Gestational Weight Gain; Anemia of Pregnancy; Stunting; Pregnancy Complications
Keywords: Pregnancy; Birth weight; Energy and protein; Micronutrients; Antenatal care; Nutrition; Birth outcomes
MeSH Terms: conditions — Fetal Growth Retardation; Premature Birth; Gestational Weight Gain; Growth Disorders; Pregnancy Complications; Birth Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1 (Active Comparator): Multiple Micronutrient Supplement for Pregnant women (UNIMMAP formulation) containing 15 nutrients all at a recommended daily allowance (RDA) for pregnancy to be consumed one-per-day during pregnancy
  Interventions: Dietary Supplement: Multiple Micronutrient Supplement for pregnant women
- Arm 2 (Experimental): Balanced energy and protein (BEP) food supplement (ready-to-use) for pregnant women containing 15 nutrients all at an RDA for pregnancy, and Ca and P. to be consumed one-per-day during pregnancy. BEP is recommended by the World Health Organization (WHO) for pregnancy use in undernourished contexts. Bangladesh is one such place. In this arm all pregnant women will receive this intervention
  Interventions: Dietary Supplement: Balanced energy and protein supplement for pregnant women
- Arm 3 (Experimental): Balanced energy and protein food supplement (ready-to-use) for pregnant women containing 15 nutrients all at an RDA for pregnancy, and Ca and P. to be consumed one-per-day during pregnancy. BEP is recommended by the WHO for pregnancy use in undernourished contexts. Bangladesh is one such place. In this arm, only low pre-pregnancy BMI women (<18.5) will receive the BEP, the rest will receive the MMS.
  Interventions: Dietary Supplement: Balanced energy and protein supplement for pregnant women
- Arm 4 (Experimental): Balanced energy and protein food supplement (ready-to-use) for pregnant women containing 15 nutrients all at an RDA for pregnancy, and Ca and P. to be consumed one-per-day during pregnancy. BEP is recommended by the WHO for pregnancy use in undernourished contexts. Bangladesh is one such place. In this arm, only low pre-pregnancy BMI women (<18.5) and those who have inadequate gestational weight gain during pregnancy will receive the BEP, the rest will receive the MMS.
  Interventions: Dietary Supplement: Balanced energy and protein supplement for pregnant women

INTERVENTIONS:
Dietary Supplement: Balanced energy and protein supplement for pregnant women — A fortified balanced energy and protein supplement providing both macro and micronutrients recommended for use during pregnancy in undernourished contexts.
  Other Names: BEP
  Arms: Arm 2; Arm 3; Arm 4
Dietary Supplement: Multiple Micronutrient Supplement for pregnant women — Prenatal supplements containing vitamins and minerals - also called "multiple micronutrient" supplements will be used in the control group.
  Other Names: MMS
  Arms: Arm 1

SUMMARY:
The primary aim of the study is to evaluate the effect of fortified balanced energy and protein (BEP) supplementation vs. control (multiple micronutrient supplement, MMS) without targeting and with targeting (either by low prepregnancy BMI or low prepregnancy BMI and inadequate gestational weight gain) on birth weight and adverse birth outcomes of low birth weight (LBW < 2500 g) and small-for-gestational age (SGA). To do this we are proposing a cluster-randomized, open labeled effectiveness trial with four arms The main question[s] it aims to answer are:

• Does mean birth weight and rate of LBW and SGA differ among mothers randomized to four arms that include targeted or untargeted BEP supplementation vs. MMS differ.

Participants will be recruited in early pregnancy and be enrolled in the trial and randomly receive:

1. A daily BEP supplement from enrollment until birth
2. A daily BEP supplement from enrollment until birth, if they have low pre-pregnancy BMI with the rest receiving a MMS supplement
3. A daily BEP supplement from enrollment until birth, if they have low pre-pregnancy BMI with the rest receiving a MMS supplement or get switched to a BEP supplement based on inadequate gestational weight gain.

Researchers will compare the above groups to women receiving a MMS daily to see if birth weight is higher in the intervention arms. Other adverse outcomes such as low birth weight, small-for-gestational age and preterm birth will also be compared between groups and relative to the control.

DETAILED DESCRIPTION:
The primary aim of the study is to evaluate the effect of a fortified balanced energy and protein (BEP) supplementation vs. control (multiple micronutrient supplement, MMS) without targeting and with targeting (either by low pre-pregnancy BMI or low pre-pregnancy BMI and inadequate gestational weight gain) on birth weight, low birth weight and SGA as the main outcomes. To do this we are proposing a cluster-randomized, open labeled effectiveness trial with four arms . Our main overall aim is:

1. To compare the mean birth weight and rates of LBW and SGA among mother randomized across four arms including targeted and untargeted BEP versus MMS.

   Additionally, to examine the effectiveness of untargeted and targeted BEP supplementation as follows:
2. To compare the mean birth weight, and rates of LBW and SGA among mothers who were randomized to receive BEP supplementation versus control (MMS) during pregnancy. [arm 2 versus 1]
3. To compare mean birth weight and rates of LBW and SGA among mothers who were randomized to receive BEP supplementation based on low pre-pregnancy BMI (w/wo inadequate gestational weight gain) versus control (MMS) during pregnancy. [arms 3+4 versus 1]
4. To compare mean birth weight and rates of LBW and SGA mothers who were randomized to receive BEP supplementation based on low pre-pregnancy BMI (w/wo inadequate gestational weight gain) versus BEP supplementation during pregnancy regardless of pre-pregnancy BMI. [arms 3+4 versus 2]

In addition to the above comparisons, between group differences and 95% confidence intervals will be estimated for both primary and secondary outcomes (shown below), with specific comparisons as described below for the primary outcome of birth weight.

Secondary Aims:

1. To compare the mean birth weight and rates of LBW and SGA among mothers who received BEP supplementation during pregnancy based on low pre-pregnancy BMI versus untargeted BEP supplementation during pregnancy [arm 3 versus 2]
2. To compare the mean birth weight and rates of LBW and SGA among mothers who received BEP supplementation during pregnancy versus BEP supplementation during pregnancy based on low pre-pregnancy BMI and gestational weight gain. [arm 4 versus 2]
3. To compare the mean birth weight and rates of LBW and SGA among mothers who received BEP supplementation during pregnancy based on pre-pregnancy BMI only versus BEP supplementation during pregnancy based on low pre-pregnancy BMI and gestational weight gain. [arm 4 versus 3]
4. To compare the difference in mean birth weights and rates of LBW and SGA among mothers who were randomized to receive BEP without targeting or with targeting relative to the control (MMS). [arm 2 versus 1 versus arm 3 and 4 versus 1]

Other objectives of the study include:

1. Assess how low mid upper arm circumference (MUAC) compares relative to low BMI in identifying women for targeting and how well MUAC change tracks with gestational weight gain change throughout pregnancy.
2. Conduct a qualitative study in the three BEP arms of the study to better understand acceptability, use, sharing and other components of adherence to BEP among women and family members and understand women's perceptions related to the screening and targeting employed in the trial.
3. Conduct a mixed methods implementation feasibility study to assess how feasible the most effective delivery approach of BEP (according to the trial findings) would be according to national and subnational stakeholders in Bangladesh.
4. Conduct a costing and cost-effectiveness analysis to compare cost of screening and cost-effectiveness of targeted vs. an untargeted supplementation approach to inform future programs.

The study design will be conducted as a cluster-randomized, unblinded trial with 4 arms among newly pregnant women. A total of 240 sectors (unit of randomization, comprising 150-200 households with women of reproductive age) will be randomized to one of the four supplementation arms, with control arm being provided a daily multiple micronutrient supplement (MMS).

Arm 1: Control - Daily MMS Arm 2: All women receive BEP Arm 3: Low BMI women receive BEP, others receive MMS Arm 4: Low BMI women receive BEP, women with inadequate gestational weight gain get switched to BEP, other receive MMS

Study Site and Participants:

The study will be conducted in the re-sized "JiVitA" (a well established field site) study area in a rural northwestern district of Bangladesh. The BEP effectiveness trial will be done among married pregnant women of reproductive age. A home-based initial census will identify all women of reproductive age living in the selected JiVitA area. We will use the JiVitA pregnancy surveillance system entailing monthly ascertainment of last menstrual period and urine-based testing among women who missed their period in the past 30 days to identify newly pregnant women for enrollment in the study. During the surveillance weight and height of the women will be assessed to calculate pre-pregnancy body mass index (BMI).

Randomization in the study will be done at a cluster level, with JIVitA sectors being used as the unit of randomization, as done in our previous studies. At pregnancy ascertainment, women will be consented for participation in the trial, and begin receiving their daily supplements as per their random allocation at the beginning of the second trimester.

Field Procedures and Data Collection

A cadre of JiVitA female staff (known as Community Health Research Workers (CHRWs), community health research workers) who are responsible for conducting the pregnancy surveillance will also be doing monthly anthropometry and distribution of the study interventions. Enrollment into the main trial will be conducted by experienced Field Interviewers (FIs), who will also be responsible for conducting a late pregnancy visit and birth assessment visits. Once a consenting pregnant woman has reached 12-14 weeks gestation, according to last menstrual period (LMP), her local CHRW will visit her monthly to distribute BEP and MMS supplements, collect compliance measurements for both, and to collect antenatal care (ANC) visit and provider history.

Information collected from the women includes: household socioeconomic status and food security using the Food & Nutrition Technical Academy (FANTA) Household Food Insecurity Access Scale (HFAIS), pregnancy history, 7-day diet recall, 28-day morbidity recall, an empowerment and agency module based on the Women's Agency Scale, a depression module adapted from the Edinburgh Postnatal Depression Scale, and anthropometry, including weight, and MUAC. Hemoglobin levels will also be assessed using a finger-prick blood draw and Hemocue machine. A late pregnancy visit will also be conducted at about 32-34 week of gestation to collect diet, morbidity, anthropometry, depression and food security information as well as to repeat Hb. A birth surveillance system will be set up for birth notification and an early visit to the home for birth assessment and anthropometry. A female interviewer (FI) will conduct the visit to collect pregnancy outcome information, infant anthropometry (length, weight, head and chest circumference) and ask a brief questionnaire on labor and delivery and measure blood pressure. One month post livebirth or stillbirth a home visit will be done to assess infant vital status and to measure maternal weight to estimate BMI.

Monitoring Supplement Adherence and Use In this effectiveness trial, supplement distribution will be done monthly. Empty food packets and MMS blister packs will be collected back and counted. A calendar to mark daily consumption will be given as an aid. After 2 weeks a phone based assessment of number of BEP packets or MMS tablets will be done as well counseling provided for any issues related to daily adherence and to encourage high compliance.

Counseling:

All women in the trial will receive counseling for antenatal care and danger signs using the behavior change communications materials developed by the Ministry of Health of Bangladesh. In addition, pamphlets for supplement benefits and use will be used for counseling. Adequate weight gain counseling using pamphlets will be done over the course of the pregnancy, across all four arms.

Sample Size:

Our sample size estimates are based on the hypothesis that either untargeted or targeted low pre-pregnancy BMI based BEP supplementation (along with MMS to women with normal BMI) will increase birth weight by 83 g and result in a relative risk reduction of 20% and 24% in SGA and LBW, respectively, compared with supplementation with MMS alone. We anticipate a total sample size of upto 2400 (600 *4 arms) live births and up to 3800 pregnant women identified through a pregnancy surveillance over 1.5 year of enrollment for the study. This is assuming a pregnancy loss of 30% and loss to follow-up of 6% and recruitment from 240 (or 60 per arm) sectors (units created in JiVitA and used for cluster randomization) across 6-8 Unions (sub-district administrative unit) of northwestern Bangladesh.

Data Analysis Our primary treatment effects analysis will be done on singleton livebirths. The analysis will be an intention-to-treat approach, i.e. all study outcomes will be analyzed as randomized. We will present crude estimates of all primary and secondary outcomes with their 95% confidence intervals adjusted for clustering at the sector level using Huber-White sandwich estimators.

ELIGIBILITY:
Inclusion Criteria:

* Married women of reproductive age (15-35 y)
* living in the selected study area who are pregnant and consent to participate in the study.

Exclusion Criteria:

* Currently pregnant or lactating women (through 12 months postpartum),
* Married women who are sterilized or widowed/divorced will not be included in the pregnancy surveillance being used to identify newly pregnant women.
* Women with gestational age of >=28 weeks of gestation using reported last menstrual period.

Ages: 15 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 3390 (Actual)
Dates: Start 2022-10-15 (Actual); Primary Completion 2025-04-23 (Actual); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Birth weight | Weight taken within 0-72 hours of birth
  Birth weight
Low birth weight (weight < 2500 g) at birth | Weight taken within 0-72 hours of birth
  Dichotomous representation of the primary outcome
Small-for-gestational age | Measured within 0-72 hours of birth
  Weight for a given gestational age lower than the 10th percentile of the reference standard

SECONDARY OUTCOMES:
Birth length | Measured within 0-72 hours of birth
  Birth length
Gestational weight change | weight from pre-pregnancy to weight measured at birth
  Gestational weight change during pregnancy
Proportion of inadequate gestational weight gain | From pre-pregnancy to birth
  Proportion of women with inadequate gestational weight gain
Head circumference at birth | at birth
  Head circumference
Chest circumference at birth | at birth
  chest circumference
Large for gestational age at birth | at birth
  Weight for gestational age > 10th percentile using fetal growth standards

OTHER OUTCOMES:
Length-for-age Z score at birth | At Birth
  Length-for-age Z score (LAZ)
weight-for-length Z score at birth | At Birth
  Weight-for-length (WLZ)
Stunting at birth | At birth
  LAZ < -2
Wasting at birth | At birth
  WLZ < -2
Short length for gestational age | At birth
  Length at birth < 10th percentile for gestational age at birth using fetal growth standards
Postpartum BMI | 1 month postpartum
  BMI at 1 month postpartum
Maternal Hemoglobin | At the third trimester (27-40 weeks)
  Maternal Hemoglobin at the third trimester
Maternal Anemia | At the third trimester (27-40 weeks)
  Maternal Anemia at the third trimester
Weight for gestational age percentile | Weight assessed within 72 hours of birth
  This is a continuous measure from which SGA using < 10th percentile (primary outcome) is defined. Uses birth measurement and gestational age at birth
Gestational blood pressure (systolic and diastolic), mmHg | During pregnancy (up to 40 weeks of gestation)
  Systolic and diastolic BP (mmHg) taken at different visits
Gestational hypertension | During pregnancy (up to 40 weeks of gestation)
  Gestational hypertension defined as high blood pressure >=140/90 mmHg that begins after 20 weeks of gestation

CONTACTS AND LOCATIONS:
Overall Officials: Parul Christian, DrPH, Principal Investigator — Johns Hopkins University
Locations (1):
- JiVitA Project, Rangpur City, Bangladesh

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data (IPD) may be shared after 2-3 years of all primary /secondary publications have appeared to the funder and researchers who request pooled analysis requiring the type of data we collect, specifically investigators who are planning to conduct similar research and testing similar interventions as ours. Data will also be shared with the funder - the Bill & Melinda Gates foundation.

REFERENCES:
- [Derived] Zavala E, Mohan D, Ali H, Siddiqua TJ, Haque R, Ayesha K, Ahsan KB, Sujan HM, Khaled N, Rahman A, Chakraborty B, Dyer B, Wu LSF, Kalbarczyk A, Erchick DJ, Thorne-Lyman AL, Tumilowicz A, Afsana K, Christian P. Targeting strategies for balanced energy and protein (BEP) supplementation in pregnancy: study protocol for the TARGET-BEP cluster-randomized controlled trial in rural Bangladesh. Trials. 2024 May 13;25(1):315. doi: 10.1186/s13063-024-08135-4. PMID 38741174